CLINICAL TRIAL: NCT07297043
Title: Efficacy of Er:YAG Laser in Removal of Impacted Mandibular Third Molars (A Randomized Controlled Clinical Trial)
Brief Title: Efficacy of Er:YAG Laser in Removing Impacted Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Karim Anwer Ahmed Nazmy, Postgraduate Researcher, Oral Laser Applications, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALEXDEN-KA-IMP_M3-2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Impacted Mandibular Third Molar
Keywords: Third Molar Surgery; Er:YAG Laser; Laser-Assisted Surgery; Oral Surgery
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned into two parallel groups: Er:YAG laser-assisted surgery and conventional rotary instrument surgery.
Masking Description: No masking was performed because both the surgeon and the participants were aware of the intervention type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:YAG Laser Group (Experimental): Participants in this group will undergo impacted mandibular third molar surgery using the Er:YAG laser for bone removal.
  Interventions: Device: Er:YAG laser
- Conventional Rotary Instrument Group (Active Comparator): Participants in this group will undergo impacted mandibular third molar surgery using conventional rotary instruments (bur and handpiece) for bone cutting.
  Interventions: Procedure: Conventional Rotary Instruments Surgery

INTERVENTIONS:
Device: Er:YAG laser — Er:YAG laser (2940 nm) used for bone cutting during impacted mandibular third molar surgery.
  Arms: Er:YAG Laser Group
Procedure: Conventional Rotary Instruments Surgery — Conventional rotary instruments used for bone removal during surgical extraction of impacted mandibular third molars.
  Arms: Conventional Rotary Instrument Group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the efficacy of the Er:YAG laser in the removal of impacted mandibular third molars compared to the conventional surgical technique. The study assesses surgical efficiency, postoperative pain, swelling, trismus, and overall patient recovery. The goal is to determine whether the Er:YAG laser provides a safer and less traumatic alternative to traditional bone-cutting methods during third molar surgery.

DETAILED DESCRIPTION:
Impacted mandibular third molars are among the most commonly extracted teeth, and conventional surgical removal often involves bone cutting using rotary instruments, which may increase postoperative morbidity. Laser-assisted surgery, particularly using the Er:YAG laser, has been proposed as a minimally invasive alternative with potential benefits such as reduced thermal damage, improved healing, and less postoperative discomfort.

This study compares Er:YAG laser-assisted bone removal with the conventional bur technique in terms of operative time, intraoperative ease, and postoperative outcomes including pain, edema, and trismus. Patients meeting the eligibility criteria are randomly allocated into two groups: a laser-assisted surgery group and a conventional surgery group. Standardized measurements and follow-up assessments are conducted to evaluate clinical outcomes and determine the effectiveness and safety of the Er:YAG laser in third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 20-30 years requiring surgical extraction of a mesioangular impacted mandibular third molar.

  * Healthy individuals with no systemic diseases that may influence bone metabolism or wound healing.
  * Good oral hygiene and absence of local infection at the surgical site.
  * No contraindications to local anesthesia, surgical extraction, or use of the Er:YAG laser.
  * Radiographic evidence confirming normal bone structure without cysts or pathological lesions.
  * Willingness to participate and ability to provide informed consent.

Exclusion Criteria:

* • Systemic medical conditions affecting bone healing or postoperative response (e.g., uncontrolled diabetes, immunodeficiency, metabolic bone disorders).

  * Current or recent use of medications influencing bone remodeling (e.g., bisphosphonates, corticosteroids, immunosuppressants).
  * Heavy smoking (>10 cigarettes/day).
  * Pregnant or breastfeeding females.
  * Poor oral hygiene, active infection, or pericoronitis at the surgical site.
  * Previous surgery, trauma, or pathology in the mandibular third molar region.
  * Known allergies or contraindications to any material or procedure used in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Immediate postoperative, 24 hours, 3 days, and 7 days
  Postoperative pain will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain) at postoperative intervals.

SECONDARY OUTCOMES:
Postoperative Swelling | Immediate postoperative, 24 hours, 3 days, and 7 days
  Facial swelling will be measured using linear facial measurements (tragus-pogonion and gonion-pogonion distances) preoperatively and at postoperative intervals.
Postoperative Trismus | Immediate postoperative, 24 hours, 3 days, and 7 days
  Maximum interincisal mouth opening will be measured in millimeters preoperatively and at postoperative intervals to assess trismus.
Bone Density | Immediate postoperative, 1 month, and 3 months
  Bone density at the extraction site will be assessed using standardized digital radiographs. Gray-scale values will be measured at predetermined reference points to compare bone healing between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Elhaw, MSc (Oral Laser Applications), Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined. Decisions regarding IPD sharing will depend on institutional policies, ethical approvals, and future publication requirements.